CLINICAL TRIAL: NCT07190820
Title: Comparison of the Accuracy of Digital and Conventional Impression in Edentulous Arch
Brief Title: Comparison of Accuracy of Full-arch Implant Digital and Conventional Impressions.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, associate professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2025-T290-1
Record Dates: First submitted 2025-08-18; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Edentulous Jaw
Keywords: digital impression; implant restoration
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital impression (Experimental)
  Interventions: Procedure: digital impression
- conventional impression (Active Comparator)
  Interventions: Procedure: conventional impression

INTERVENTIONS:
Procedure: digital impression — complete arch implant impression with intraoral photogrammetry
  Arms: digital impression
Procedure: conventional impression — conventional open tray splint impression
  Arms: conventional impression

SUMMARY:
The goal of this clinical trial is to determine whether the accuracy of digital impressions is comparable to conventional impressions. It will also learn about the clinical effect of different method. The main questions it aims to answer are: Does drug ABC lower the number of times participants need to use a rescue inhaler? What medical problems do participants have when taking drug ABC? Researchers will compare digital impression to conventional impression to see if the accuracy of the digital method.

Participants will:

Take an impression with one of the methods Visit the clinic a total of 6 times for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-80 years (inclusive) with no gender restriction.
* Patients who will receive a full-arch one-piece implant-supported fixed
* permanent restoration in the maxilla or mandible.
* Patients with osseointegrated implants after surgery.
* Patients voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Patients with a severe gag reflex.
* Patients with insufficient interarch space in the posterior region for impression coping placement.
* Patients with minimal inter-implant distance may prevent impression coping installation.
* Patients with temporomandibular joint (TMJ) disorders are unable to maintain prolonged mouth opening for impression procedures.
* Other conditions deemed ineligible for inclusion by the investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vision and tactile score for evaluating passive fit of metal framework | Periprocedural: At the time of the titanium framework try-in: the try-in of the framework to the patient is before final delivery. (The delivery of the final prosthesis is the baseline)
  Five aspects are evaluated, each aspect is scored as 0 or1. The score ranges from 0 to 5 points. 1、Framework rocking upon seating？2、 Gap assessment with single screw test. The method utilized an explorer with an approximately Ø60-µm tip to evaluate the margins of the metal framework.3、 Gap assessment with all screws tightened. 4、Are the screws threading smoothly? 5、Radiographic assessment of framework fit (check for gaps).

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT07190820/Prot_SAP_000.pdf